CLINICAL TRIAL: NCT07341750
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of Bacillus Coagulans SNZ 1969 on Immune Health in Healthy School-aged Children
Brief Title: Effects of Bacillus Coagulans SNZ 1969 on Immune Health in Healthy School-aged Children
Acronym: BC SNZ 1969
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanzyme Biologics Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25SACCP01; 79156228 (Other: ISRCTN, UK clinical trials registry)
Record Dates: First submitted 2025-11-25; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Immunity
Keywords: Probiotic immune health; Bacillus coagulans; Bacillus coagulans SNZ 1969

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Bacillus coagulans SNZ 1969 arm (Active Comparator): Bacillus coagulans SNZ 1969 sachet containing 1 Billion CFU/g.
  Interventions: Dietary Supplement: Probiotic formulation
- Placebo arm (Placebo Comparator): Placebo Ingredients: Glucidex (Maltodextrin), Magnesium Stearate, Banana dry mix flavour.
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Probiotic formulation — Bacillus coagulans SNZ 1969 1 Billion CFU/g in sachet form with non-medicinal ingredients: Glucidex (maltodextrin), Magnesium stearate, Banana dry mix flavour. Participants will be instructed to fully consume 1 sachet containing 1 Billion CFU/g completely dissolved in approximately 50 ml of water before breakfast starting on Day 1 and throughout the duration of the study.
  Arms: Probiotic Bacillus coagulans SNZ 1969 arm
Dietary Supplement: Placebo Control — Placebo Ingredients: Glucidex (Maltodextrin), Magnesium Stearate, Banana dry mix flavour. Participants will be instructed to fully consume 1 sachet completely dissolved in approximately 50 ml of water before breakfast starting on Day 1 and throughout the duration of the study.
  Arms: Placebo arm

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of Bacillus coagulans SNZ 1969 on immune health in healthy school-aged children in terms of reduction of respiratory symptoms, gastrointestinal symptoms, immunoglobulins, immune biomarkers and fecal microbiome changes.

The current study will examine the efficacy of Bacillus coagulans SNZ 1969 (B. coagulans) on immune health in children attending school. The primary outcome will assess the difference between the investigational product and placebo from baseline to day 84 in incidence, duration, and severity of Upper Respiratory Tract Infection (URTI) and Gastrointestinal Tract Infection (GITI) symptoms. This will be assessed by use of the Canadian Acute Respiratory Illness and Flu Scale (CARIFS) and a GITI symptoms questionnaire.

Enrolled participants will include children 6-12 years of age currently attending school during the 2025-2026 cold and flu season to allow for adequate exposure to URTI or GITI pathogens. To avoid confounding effects of pre-existing medical conditions children presenting with a history or presence of a clinically relevant respiratory, pulmonary, or gastrointestinal condition will be excluded at the discretion of the Qualified Investigator. Furthermore, participants consuming immune modulating medications, antibiotics, products containing B. coagulans, or any other probiotic supplement will be excluded unless they have undergone the specified washout. The strict eligibility criteria is designed to reduce confounders on immune health affecting both upper respiratory tract infections and gastrointestinal tract infection symptoms. Children presenting with any other medical condition or lifestyle factor which may affect the safety of their participation or study outcomes will also be excluded.

Each participant will be assigned a randomization code according to the order of the randomization list generated. Enrolled participants will be randomized to the different study arms at Day 0. Participants will take either probiotic Bacillus coagulans SNZ 1969 or a placebo every day for 84 days.

Day 0 (Baseline, Visit 2) Eligible volunteers will return to the clinic for baseline assessments with collected stool and saliva samples.

Baseline (Day 0) assessments include:

1. Review concomitant therapies (inclusive of previous vaccinations) and current health status
2. Assess inclusion and exclusion criteria
3. Review any pre-emergent AEs
4. Urine pregnancy test for potential volunteers that are of child-bearing potential
5. Vital sign measurements (BP and HR)
6. Weight and height measurements
7. Randomization of eligible participants
8. Collect blood samples for analysis of:

   1. Quantibody® Human Immune Response Array
   2. Immunoglobulins A (IgA), G (IgG), E (IgE) and M (IgM) serum levels
9. Collect saliva sample for the analysis of Salivary Ig A Levels
10. Collect stool samples for microbiome analysis
11. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
12. Dispense investigational product and instruct participants on use
13. Dispense study diary inclusive of the CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
14. Dispense stool collection kit for microbiome analysis for Visit 5 (End of Study visit)
15. Dispense saliva collection kit for Visit 5 (End of Study visit) The next visit will be conducted remotely and scheduled for Day 28 (± 2 days) and Day 56 (± 2 days).

End of Study (Day 84 ± 2 days):

Participants will return to the clinic for end of study assessments, with unused investigational product, completed study diaries (inclusive of the CARIFs, Additional respiratory tract symptoms, and GITI symptoms questionnaires), and stool and saliva samples.

Visit 5 assessments include:

1. Return and review study diary
2. Return unused investigational product in the original packaging and remnants and calculate compliance by counting the returned unused investigational product
3. Review concomitant therapies and AEs
4. Vital sign measurements (BP and HR)
5. Weight and height measurements
6. Urine pregnancy test for participants that are of childbearing potential
7. Collect blood samples for the analysis of:

   1. Quantibody® Human Immune Response Array
   2. Immunoglobulins A (IgA), G (IgG), E (IgE) and M (IgM) serum levels
8. Collect saliva samples for the analysis of Salivary Ig A Levels
9. Collect stool samples for microbiome analysis
10. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires

DETAILED DESCRIPTION:
The current study will examine the efficacy of Bacillus coagulans SNZ 1969 (B. coagulans) on immune health in children attending school. The primary outcome will assess the difference between the investigational product and placebo from baseline to day 84 in incidence, duration, and severity of Upper Respiratory Tract Infection (URTI) and Gastrointestinal Tract Infection (GITI) symptoms. This will be assessed by use of the Canadian Acute Respiratory Illness and Flu Scale (CARIFS) and a GITI symptoms questionnaire. Enrolled participants will include children 6-12 years of age currently attending school during the 2025-2026 cold and flu season to allow for adequate exposure to URTI or GITI pathogens. To avoid confounding effects of pre-existing medical conditions children presenting with a history or presence of a clinically relevant respiratory, pulmonary, or gastrointestinal condition will be excluded at the discretion of the Qualified Investigator. Furthermore, participants consuming immune modulating medications, antibiotics, products containing B. coagulans, or any other probiotic supplement will be excluded unless they have undergone the specified washout. The strict eligibility criteria is designed to reduce confounders on immune health affecting both upper respiratory tract infections and gastrointestinal tract infection symptoms.

Children presenting with any other medical condition or lifestyle factor which may affect the safety of their participation or study outcomes will also be excluded. The planned sample size for this study is 100. In order to evaluate primary, secondary, and safety outcomes, study assessments will be conducted as per the Schedule of Assessments.

Screening (Day -45 to Day -15; Visit 1)*

* At the discretion of the Qualified Investigator, any participants falling outside of the screening window (Day -45 to Day -15) due to scheduling issues will be asked to repeat eligibility/screening procedures prior to randomization at baseline.

At screening, an ICF will be given to the potential volunteer. They will be required to read the information and will be given the opportunity to seek more information if needed or provided with the option of taking the consent form home to review prior to making their decision. If agreeable, the caregiver and volunteer will sign the consent and assent forms as applicable and receive a duplicate of the signed copy. Once consent has been obtained, screening will proceed. Each volunteer will be assigned a screening number to be entered in the screening and enrollment log.

Screening assessments include:

1. Review medical history, concomitant therapies (inclusive of previous vaccinations), and current health status
2. Assess inclusion and exclusion criteria
3. Review any pre-emergent AEs
4. Urine pregnancy test for potential volunteers that are of child-bearing potential
5. Seated resting BP and HR measurements
6. Weight and height measurements
7. Dispense study diary inclusive of the CARIFS questionnaire, Additional respiratory tract symptoms questionnaire, and GITI Symptom Questionnaire and instruct participants on completion
8. Dispense saliva collection kit and instruct participants on use
9. Dispense stool collection kit and instruct participants on use The next appointment will be scheduled for potentially eligible volunteers for their baseline visit.

Run-in (Day -14 to Day -1):

Participants will complete the study diary inclusive of the CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires during the 14-day run-in period.

Day 0 (Baseline, Visit 2):

Eligible volunteers will return to the clinic for baseline assessments with collected stool and saliva samples.

Baseline (Day 0) assessments include:

1. Review concomitant therapies (inclusive of previous vaccinations) and current health status
2. Assess inclusion and exclusion criteria
3. Review any pre-emergent AEs
4. Urine pregnancy test for potential volunteers that are of child-bearing potential
5. Vital sign measurements (BP and HR)
6. Weight and height measurements
7. Randomization of eligible participants
8. Collect blood samples for analysis of:

   1. Quantibody® Human Immune Response Array
   2. Immunoglobulins A (IgA), G (IgG), E (IgE) and M (IgM) serum levels
9. Collect saliva sample for the analysis of Salivary Ig A Levels
10. Collect stool samples for microbiome analysis
11. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
12. Dispense investigational product and instruct participants on use
13. Dispense study diary inclusive of the CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
14. Dispense stool collection kit for microbiome analysis for Visit 5 (End of Study visit)
15. Dispense saliva collection kit for Visit 5 (End of Study visit) The next visit will be conducted remotely and scheduled for Day 28 (± 2 days) Visit 3 (Day 28 ± 2 days) Participants will attend remotely for Visit 3 assessments with completed study diaries inclusive of the CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires.

Visit 3 assessments include:

1. Review compliance by referencing study diaries and participant/caregiver count of study product
2. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
3. Review concomitant therapies and AEs
4. Dispense new study diary The next visit will be conducted remotely and scheduled for Day 56 (± 2 days). Visit 4 (Day 56 ± 2 days) Participants will attend remotely for Visit 4 assessments with completed study diaries inclusive of the CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires.

Visit 4 assessments include:

1. Review compliance by referencing study diaries and participant/caregiver count of study product.
2. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires
3. Review concomitant therapies and AEs
4. Dispense new study diary
5. Participants will be reminded to bring saliva and stool samples for the End of Study visit.

The next visit will be scheduled for Day 84 (± 2 days). Visit 5 - End of Study (Day 84 ± 2 days) Participants will return to the clinic for end of study assessments, with unused investigational product, completed study diaries (inclusive of the CARIFs, Additional respiratory tract symptoms, and GITI symptoms questionnaires), and stool and saliva samples.

Visit 5 assessments include:

1. Return and review study diary
2. Return unused investigational product in the original packaging and remnants and calculate compliance by counting the returned unused investigational product
3. Review concomitant therapies and AEs
4. Vital sign measurements (BP and HR)
5. Weight and height measurements
6. Urine pregnancy test for participants that are of childbearing potential
7. Collect blood samples for the analysis of:

   1. Quantibody® Human Immune Response Array
   2. Immunoglobulins A (IgA), G (IgG), E (IgE) and M (IgM) serum levels
8. Collect saliva samples for the analysis of Salivary Ig A Levels
9. Collect stool samples for microbiome analysis
10. Review completed study diaries including CARIFS, Additional respiratory tract symptoms, and GITI symptoms questionnaires.

This study will be conducted with the highest respect for the individual participants (i.e., participants) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the ICH Harmonised Tripartite Guideline for GCP. Written consent documents will embody the elements of informed consent as described in the declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all applicable laws and regulations. The ICF describes the planned and permitted uses, transfers, and disclosures of the volunteer's personal and personal health information for purposes of conducting the study. The ICF further explains the nature of the study, its objectives, and potential risks and benefits, as well as the date informed consent is obtained. The ICF will detail the requirements of the volunteer and the fact that he or she is free to withdraw at any time without giving a reason and without prejudice to his or her further medical care.

Study monitoring:

Source documents will be reviewed to ensure that all items have been completed and that the data provided are accurate and obtained in the manner specified in the protocol. The participant files will be reviewed to confirm that:

1. Informed consent was obtained and documented
2. Enrolled participants fulfilled all inclusion criteria and did not meet any exclusion criteria;
3. AE/SAE reporting has been performed as applicable
4. Study visits have been conducted as per protocol and information has been recorded in the appropriate place in the source document
5. The study product is being stored correctly and an accurate record of its dispensation to the study participants is being maintained (accountability) Incorrect, inappropriate, or illegible entries in the participant files will be returned to the Qualified Investigator or designee for correction. No data disclosing the identity of participants will leave the study center. The Qualified Investigator and any designees will maintain confidentiality of all participant records.

The Qualified Investigator will permit study-related monitoring, audits, IRB/IEC review, and regulatory inspections and will allow direct access to source data and documents for these purposes. Data required for the analysis will be acquired from source documentation (including laboratory reports) and captured through electronic data capture (EDC) case report forms specifically designed for this study.

A password-protected user ID is created giving access to the delegated study personnel. The data management personnel designs the database, and once the database is finalized study-specific Data Management Plan is generated.

The standard data validation and edit checks are performed by designing study-specific rules and restrictions defined in the eCRF. The discrepancies will be queried and managed. Data sets will be created, queried, and exported during and at the end of the study.For Statistical analysis, the data management personnel provides a validated locked blinded database to the Statistician to perform the analysis.

High safety standards for the transfer and storage of study data are guaranteed by the use of technologies such as password protection, firewalls, and periodic backup to protect stored data. All study data is archived for a period not less than 15 years from the date of completion of the study in accordance with Health Canada regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 6 and 12 years of age at screening, inclusive.
* Children enrolled in and attending school in person at baseline.
* Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic and remote visits.
* A care provider who can reliably bring the participant to study visits. The participant's primary caregiver must be willing and able to complete the questionnaires.
* The participant or the participant's parents/guardian are willing and able to provide written assent and/or informed consent as appropriate.
* Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study.
* Healthy as determined by medical history as assessed by the Qualified Investigator (QI).

Exclusion Criteria:

* Individuals who are pregnant.
* Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of the investigational product or placebo ingredients.
* History or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), respiratory, pulmonary, biliary, metabolic, haematologic, gastrointestinal, or pancreatic disorders, that may affect participation or outcomes as assessed by the QI.
* Confirmed history of COVID-19 infection in the 3 months prior to baseline.
* Immune dysfunction, autoimmune disease, immune compromised and/or taking an immunosuppressive medication, as assessed by the QI.
* Severe environmental allergies requiring medical or need for allergy shots, as assessed by the QI.
* Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI.
* Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable.
* Asthma, as assessed by the QI.
* Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and or safety of the investigational product.
* Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI.
* Participant or participant's caregiver who are cognitively or neurodevelopmentally impaired affecting their ability to give informed consent and/or assent.
* Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
URTI SYMPTOMS | baseline to day 84
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of URTI as assessed by the Canadian Acute Respiratory Illness and Flu Scale (CARIFS) from baseline to day 84 between Bacillus coagulans SNZ 1969 and Placebo. CARIFS Scoring: 18 items, each scored 0 (none) to 3 (severe), yielding a total score from 0 to 54 (higher score = worse illness).
ADDITIONAL RESPIRATORY TRACT SYMPTOMS | baseline to day 84
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of Additional Respiratory Tract Symptoms as assessed by Additional Respiratory Tract Symptoms questionnare from baseline to day 84 between Bacillus coagulans SNZ 1969 and placebo. Additional Respiratory Tract symptoms Scale: Usually 0 (None) to 3 (Severe) with higher scores indicating greater severity.
GITI symptoms | baseline to day 84
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of GITI symptoms as assessed by the GITI Symptoms Questionnaire from baseline to day 84 between Bacillus coagulans SNZ 1969 and placebo. GITI Symptom questionnaire is rated on a three-point Likert-type scale ranging from 0 to 2, with a higher score signifying more severe GI symptoms.

SECONDARY OUTCOMES:
Canadian Acute Respiratory Illness and Flu Scale (CARIFS) | baseline to days 28 and 56
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of URTI as assessed by the CARIFS from baseline to days 28 and 56 between B coagulans SNZ 1969 and placebo. CARIFS Scoring: 18 items, each scored 0 (none) to 3 (severe), yielding a total score from 0 to 54 (higher score = worse illness).
Additional Respiratory tract symptoms | Baseline to days 28 and 56
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of Additional Respiratory tract symptoms as assessed by Additional Respiratory Tract Symptoms questionnare from baseline to days 28 and 56 between B coagulans SNZ 1969 and placebo. Additional Respiratory Tract symptoms Scale: Usually 0 (None) to 3 (Severe) with higher scores indicating greater severity.
GITI Symptoms | Baseline to days 28 and 56
  The difference in incidence - Proportion (%), duration - days, and severity (area-under-the-curve (AUC) - score days) of GITI symptoms as assessed by the GITI Symptoms Questionnaire from baseline to days 28 and 56 between B. coagulans SNZ 1969 and placebo. GITI Symptom questionnaire is rated on a three-point Likert-type scale ranging from 0 to 2, with a higher score signifying more severe GI symptoms.
Total and individual daily symptoms | baseline to days 28, 56, and 84
  The difference between B. coagulans SNZ 1969 and placebo on the severity of cold/flu and GITI symptoms as assessed by total and individual daily symptoms
Missed school days | baseline to days 28, 56, and 84
  The difference between B. coagulans SNZ 1969 and placebo on the number of missed school days
Number of well days | baseline to days 28, 56, and 84
  The difference between B. coagulans SNZ 1969 and placebo from on the number of well days, related to the absence of cold/flu and GITI symptoms
Use of cold/flu medications | baseline to days 28, 56, and 84
  The difference between B. coagulans SNZ 1969 and placebo on the use of prescription and non-prescription cold/flu medications to treat cold or flu symptoms
Total days of illness | baseline to days 28, 56, and 84
  The difference between B. coagulans SNZ 1969 and placebo on the total days of illness

OTHER OUTCOMES:
Immunoglobulins | Baseline to day 84
  Saliva secretory immunoglobulin A (sIgA) concentrations; Serum levels of Immunoglobulin A (IgA), G (IgG), E (IgE) and M (IgM)
Immune response biomarkers | baseline to day 84
  Immune related protein serum levels (pg/mL) of - CD14, CD163, CD40 (TNFRSF5), CRP (C-Reactive Protein), E-Selectin, Fas (TNFRSF6/Apo-1), Fas Ligand (TNFSF6), GCSF, ICAM-1 (CD54), IL-1 alpha (IL-1 F1), IL-1 beta (IL-1 F2), IL-1 R4 (ST2), IL-10, IL-12 p70, IL-13, IL18, IL-2, IL-2 R alpha, IL-4, IL-6, IL-8 (CXCL8), Lipocalin-2 (NGAL), MCP-1 (CCL2), MCP-2 (CCL8), MIF, MIP-1 alpha (CCL3), MIP-1 beta (CCL4), Osteopontin (SPP1), PAI-1, Platelet Factor 4 (CXCL4), Procalcitonin, RAGE, Resistin, Thrombomodulin, TNF alpha, TREM-1, Troponin I, uPAR, VCAM-1 (CD106), VEGF-A. The units of measurement for all the Immune Biomarkers are in pg/mL).
Fecal microbiome analysis | baseline to day 84
  Microbiome as assessed by 16s rRNA fecal microbiome analysis
Safety and Tolerability - Incidence of post-emergent adverse events (AE). | through study completion upto Day 84
  Number of participants with Incidence of post-emergent adverse events (AE)
Changes in Vital signs (Blood Pressure) | through study completion upto Day 84
  Number of participants with clinically relevant changes in vital signs - Blood Pressure [Systolic blood pressure (SBP)/Diastolic blood pressure (DBP)] with units in millimeters of mercury (mmHg) after supplementation
Changes in Vital signs (Heart Rate) | through study completion upto Day 84
  Number of participants with clinically relevant changes in vital signs - Heart rate (HR) with units in bpm (beats per minute) after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc. 275 Dundas Street, Tower A Suite G025 London, ON N6B 3L1 Canada, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No